CLINICAL TRIAL: NCT03199157
Title: The Effect Of Fentanyl 12 Mcg Transdermal Patch On Postoperative Pain Following Unilateral, Single-Level Laminectomy/Discectomy: A Randomized, Controlled, Double-Blind Study
Brief Title: Fentanyl 12 Mcg Transdermal Patch For Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Oya Yalcin Cok, Medical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA14-66
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl Group (Active Comparator): Patients received the fentanyl 12 mcg transdermal patch (FG, n=38) 8 hours preoperatively and until 24 hours after the surgery
  Interventions: Drug: Fentanyl transdermal patch
- Control group (No Intervention)

INTERVENTIONS:
Drug: Fentanyl transdermal patch — Patients received fentanyl 12 mcg transdermal patch group 8 hours preoperatively and until 24 hours after the surgery
  Arms: Fentanyl Group

SUMMARY:
The investigators designed a prospective randomized study to investigate the effect of fentanyl 12 mcg transdermal patch on postoperative pain following unilateral, single-level laminectomy/discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 20-70 years
* ASA physical status 1-2 patients undergoing single-level laminectomy/discectomy

Exclusion Criteria:

* A history of allergy to any study drugs
* History of opioid use, obstructive sleep apnea
* Any psychological disorders
* hepatic or renal failure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Numeric rating score for pain (NRS) | Postoperative 24 hours